CLINICAL TRIAL: NCT05822453
Title: Gemcitabine Plus S1 and Tislelizumab in the First Line Therapy of Advanced Biliary Tract Carcinoma (BTC): a Single Arm, Prospective, Interventional Clinical Study
Brief Title: Gemcitabine Plus S1 and Tislelizumab in the First Line Therapy of Advanced Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-001
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — Gemcitabine; S 1 (combination); tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine plus S1 and tislelizumab (Experimental): Participants will receive gemcitabine plus S1 and tislelizumab until disease progression or unacceptable toxicity
  Interventions: Drug: Gemcitabine; Drug: S1; Drug: Tislelizumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine (1000 mg/m2) will be administered by IV infusion on Day 1and Day 8 of each 21-day cycle
Drug: S1 — S1 (60 mg/day if body surface area < 1.25 m2, 80 mg/day if body surface area = 1.25~1.50 m2) will be administered by PO on Day 1 ~ 14 of each 21-day cycle
Drug: Tislelizumab — Tislelizumab (200 mg) will be administered by IV infusion on Day 1 of each 21-day cycle

SUMMARY:
This study will evaluate the efficacy and safety of 1st line therapy with gemcitabine plus S1 and tislelizumab in participants with advanced biliary tract carcinoma (BTC).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≤ 18 years old ≤ 75 years old, regardless of gender.
* 2. Diagnosed as malignant tumor of biliary tract by histopathology or cytology, including intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, common bile duct carcinoma or gallbladder carcinoma.
* 3. The disease is not suitable for radical surgery and/or local treatment;
* 4. At least one measurable lesion according to RECIST 1.1 standard
* 5. The ECOG score is 0-1
* 6. The expected survival ≥ 12 weeks.
* 7. The Child-Pugh score is 5-7
* 8. Within the past 2 years, there was no active autoimmune diseases that require systemic treatment, replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction)
* 9. Women with fertility: agree to abstain during treatment and at least 6 months after the last dose (to avoid heterosexual intercourse) or use contraceptive methods with an annual contraceptive failure rate of less than 1%.
* 10. Male: Agree to abstain (not engage in heterosexual intercourse) or use contraception, agree not to donate sperm
* 11. The subjects voluntarily participated in the study and agreed to sign written informed consent, with good compliance and cooperation in follow-up.

Exclusion Criteria:

* 1. who have any of the following: (1) suitable for surgical radical treatment, (2) have undergone radical surgery without assessable lesions, (3) have received first-line systemic treatment
* 2. Known to be allergic or intolerant to recombinant humanized PD-1 monoclonal antibody drugs and their components.
* 3. ECOG PS ≥ 2
* 4. metastasis site>2 organs
* 5. Pregnant or lactating women
* 6. Received local anti-tumor therapy within 4 weeks prior to the first study drug treatment, including but not limited to radiotherapy, radiofrequency ablation, cryoablation, or percutaneous ethanol injection
* 7. Receiving approved or developing systemic anticancer therapies, including chemotherapy, biological immunotherapy, targeted therapy, or Chinese herbal therapy with clear indications for anti-tumor effects
* 8. There are multiple factors that can affect the oral administration of S1 (such as inability to swallow, chronic diarrhea, intestinal obstruction, or other conditions that significantly affect drug administration and absorption)
* 9. Simultaneously participating in another clinical study
* 10. After comprehensive assessment of the condition by the investigators, it is deemed unsuitable to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline up to approximately 6 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | baseline up to approximately 12 months
1-year survival rate | baseline up to approximately 12 months
Disease control rate (DCR) | baseline up to approximately 6 months
Duration of response (DoR) | baseline up to approximately 12 months
Percentage of participants with SD ≥ 4 weeks | baseline up to approximately 6 months
3-month progression free survival rate | baseline up to approximately 3 months
6-month progression free survival rate | baseline up to approximately 6 months
6-month overall survival rate | baseline up to approximately 6 months
12-month overall survival rate | baseline up to approximately 12 months
Quality of life (QoL) | baseline up to approximately 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, China